CLINICAL TRIAL: NCT01613547
Title: The Effect of Routine Antibiotic Use in the Outpatient Treatment of Severely Malnourished Children Without Complications: Maradi, Niger
Brief Title: The Effect of Routine Antibiotic Use in the Outpatient Treatment of Severely Malnourished Children Without Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); FORSANI (Unknown); District Sanitaire de Madarounfa, Région de Maradi (Unknown); Ministere de la Sante Publique du Niger (Unknown); Bichat Hospital (Other)
Responsible Party: Principal Investigator, Sheila Isanaka, Prinicipal Investigator, Epicentre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPI/NIGER/821242
Record Dates: First submitted 2012-05-26; First posted 2012-06-07 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine antibiotic prescription (Active Comparator): Routine antibiotic prescription with amoxicillin (80 mg/kg/day for 7 days)
  Interventions: Drug: Amoxicillin
- No routine antibiotic prescription (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin — 80 mg/kg/day for 7 days
  Arms: Routine antibiotic prescription
Drug: Placebo — 7 days
  Arms: No routine antibiotic prescription

SUMMARY:
This study will be conducted as a randomized, double-blind, placebo-controlled trial to compare routine antibiotic prescription vs. no routine antibiotic prescription in the management of uncomplicated cases of severe acute malnutrition treated in the community in terms of nutritional recovery. The investigators hypothesize that there will be no significant difference in terms of the risk of nutritional recovery among children uncomplicated cases of severe acute malnutrition treated in the community that receive routine antibiotic prescription and those who receive no routine antibiotic prescription.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 59 months
* MUAC < 11.5 cm or WHZ < -3
* Absence of bipedal edema
* Absence of current illness requiring inpatient care
* Eligible for new admission for outpatient nutritional therapy for SAM at 3 CRENAS in Madarounfa operated by FORSANI
* Absence of current clinical illness requiring prescription of specific antibiotic therapy and decision by the study physician to use a specific antimicrobial drug on admission
* Written consent of parent or caregiver
* Residence within Niger

Exclusion Criteria:

* Age < 6 months or > 59 months
* MUAC ≥ 11.5 cm and WHZ ≥ -3
* Presence of bipedal edema
* Presence of current illness requiring inpatient care
* Decision by the study physician to use a specific different antimicrobial drug on admission
* Presence of any congenital abnormality or underlying chronic disease that may affect growth or risk of infection
* Treatment with any antibiotic within 7 days
* Admission to any nutritional program for the treatment of SAM within 3 months
* Known contraindication / hypersensitivity to amoxicillin

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2412 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proportion of children discharged from nutritional program as recovered | Until discharge from the nutritional program, an expected average of 5 weeks

SECONDARY OUTCOMES:
Hospitalization or death | 3 months following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Isanaka, ScD, Principal Investigator — Epicentre
Locations (1):
- Centres de Récupération et d'Education Nutritionnelle Ambulatoires de Dan Issa, Madarounfa, and Gabi, Maradi, Niger

REFERENCES:
- [Derived] Rattigan SM, Grantz KH, Hanson K, Langendorf C, Berthe F, Grais R, Isanaka S. Prescribing practices in the treatment of wasting: secondary analysis from a randomised trial. BMJ Nutr Prev Health. 2024 Feb 26;7(1):103-111. doi: 10.1136/bmjnph-2023-000785. eCollection 2024. PMID 38966095
- [Derived] Schwartz DJ, Langdon A, Sun X, Langendorf C, Berthe F, Grais RF, Trehan I, Isanaka S, Dantas G. Effect of amoxicillin on the gut microbiome of children with severe acute malnutrition in Madarounfa, Niger: a retrospective metagenomic analysis of a placebo-controlled trial. Lancet Microbe. 2023 Nov;4(11):e931-e942. doi: 10.1016/S2666-5247(23)00213-6. Epub 2023 Oct 19. PMID 37866373
- [Derived] Bliznashka L, Grantz KH, Botton J, Berthe F, Garba S, Hanson KE, Grais RF, Isanaka S. Burden and risk factors for relapse following successful treatment of uncomplicated severe acute malnutrition in young children: Secondary analysis from a randomised trial in Niger. Matern Child Nutr. 2022 Oct;18(4):e13400. doi: 10.1111/mcn.13400. Epub 2022 Jul 21. PMID 35866201
- [Derived] Madzorera I, Duggan C, Berthe F, Grais RF, Isanaka S. The role of dietary diversity in the response to treatment of uncomplicated severe acute malnutrition among children in Niger: a prospective study. BMC Nutr. 2018 Sep 20;4:35. doi: 10.1186/s40795-018-0242-y. eCollection 2018. PMID 32153896
- [Derived] Maataoui N, Langendorf C, Berthe F, Bayjanov JR, van Schaik W, Isanaka S, Grais RF, Clermont O, Andremont A, Armand-Lefevre L, Woerther PL. Increased risk of acquisition and transmission of ESBL-producing Enterobacteriaceae in malnourished children exposed to amoxicillin. J Antimicrob Chemother. 2020 Mar 1;75(3):709-717. doi: 10.1093/jac/dkz487. PMID 31821452
- [Derived] Oldenburg CE, Guerin PJ, Berthe F, Grais RF, Isanaka S. Malaria and Nutritional Status Among Children With Severe Acute Malnutrition in Niger: A Prospective Cohort Study. Clin Infect Dis. 2018 Sep 14;67(7):1027-1034. doi: 10.1093/cid/ciy207. PMID 29522089
- [Derived] Isanaka S, Langendorf C, Berthe F, Gnegne S, Li N, Ousmane N, Harouna S, Hassane H, Schaefer M, Adehossi E, Grais RF. Routine Amoxicillin for Uncomplicated Severe Acute Malnutrition in Children. N Engl J Med. 2016 Feb 4;374(5):444-53. doi: 10.1056/NEJMoa1507024. PMID 26840134